CLINICAL TRIAL: NCT04374188
Title: Efficacy of Ciprofloxacin Therapy in Avoidance of Sepsis in Patient Undergoing Percutanous Nephrolithotomy: A Randomized Controlled Trial
Brief Title: Efficacy of Ciprofloxacin Therapy in Avoidance of Sepsis in Patient Undergoing Percutanous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diaa Eldin Taha Ramadan Mohamed (Other)
Responsible Party: Sponsor-Investigator, Diaa Eldin Taha Ramadan Mohamed, Lecturer of urology, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS/19.23
Record Dates: First submitted 2020-04-18; First posted 2020-05-05 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Ciprofloxacin; Quinolones; Levofloxacin

STUDY DESIGN:
Intervention Model Description: Efficacy of ciprofloxacin therapy in sepsis avoidance.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ciprofloxacin (Active Comparator): ciprofloxacin tablets
  Interventions: Drug: Ciprofloxacin
- levofloxacin (Active Comparator): levofloxacin tablets
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — drug adminstration to ameliorate sepsis incidence
  Other Names: quinolones
  Arms: ciprofloxacin
Drug: Levofloxacin — levofloxacin pill
  Other Names: quinolones
  Arms: levofloxacin

SUMMARY:
Efficacy of ciprofloxacin therapy in avoidance of sepsis in patient undergoing percutanous nephrolithotomy. A randomized controlled trial.

DETAILED DESCRIPTION:
To figure out the value of oral ciprofloxacin medication in ameliorate the outcome of renal nephrolithiasis extraction via the endoscope as regard the sepsis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient 18 years or older
* Stones ≥ 2 cm and/or mild to moderate hydronephrosis
* Sterile mid urine stream

Exclusion Criteria:

* Patients with a stent, nephrostomy tube or indwelling catheter
* Renal failure
* Fever before surgery
* Previous manipulation/procedure
* Concomitant bladder stone or tumour
* Patients with active UTI
* Contralateral renal/ureteric stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect of ciprofloxacin versus levofloxacin duration before PCNL | 12 months
  To evaluate whether 7 days of ciprofloxacin or levofloxacin before PCNL, can reduce upper urinary tract infection and urosepsis after PCNL.

SECONDARY OUTCOMES:
differences between Culture and sensitivity (C&S) of Preoperative urine (MSU) and intraoperative renal pelvic urine | 12 months
  Compare the difference between C&S of Preoperative urine (MSU) and intraoperative renal pelvic urine and extracted stone, in predicting the upper urinary tract infection and urosepsis.
predictors of systemic inflammatory response syndeome (SIRS) and sepsis post PCNL. | 12 months
  assess the risk factors for SIRS and sepsis in PCNL.

CONTACTS AND LOCATIONS:
Overall Officials: Diaa Eldin Taha, MD, Principal Investigator — Lecturer of urology
Locations (1):
- Kafrelsheikh faculty of medicine, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No